CLINICAL TRIAL: NCT05825508
Title: PedBot Ankle Rehabilitation
Brief Title: PedBot Ankle Rehablitation
Status: Active, not recruiting | Type: Observational
Sponsor: Children's National Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00013680
Record Dates: First submitted 2023-04-11; First posted 2023-04-24 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: ankle robot — home ankle robot and video game

SUMMARY:
The primary objective of the study is to determine engagement with use and adherence to a home exercise program with our PedBotHome ankle rehabilitation device. We will place the device in the home for 90 days and consider the study a success if used for at least 30 minutes a day for at least 3 days a week during this period.

DETAILED DESCRIPTION:
The major secondary objective is to determine if the range of motion of the ankle has improved through use of PedBotHome. Other secondary objectives will measure ankle strength and control.

Secondary outcomes will include a measurable increase in range of motion across the ankle joint (in any direction) and a measurable increase in strength in plantarflexion, dorsiflexion, inversion, and eversion. Improvement in gait and speed of ambulation will also be considered secondary outcome measures as an indication of better ankle control.

ELIGIBILITY:
Inclusion Criteria:

* Cerebral palsy

Exclusion Criteria:

* Healthy volunteers

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients treated by Physical Medicine and Rehab with cerebral palsy
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-07-28 (Actual); Primary Completion 2025-07-28 (Estimated); Study Completion 2025-07-28 (Estimated)

PRIMARY OUTCOMES:
number of days used | 90 days
  integer

CONTACTS AND LOCATIONS:
Locations (1):
- Children's National Health System, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No